CLINICAL TRIAL: NCT03161275
Title: Measurement of the Cerebral Saturation for Assessment of Safety of Epidural Anaesthesia During Abdominal Surgery
Status: Completed | Type: Observational
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Tomasz Skladzien, Ph.D., Jagiellonian University
Other Study IDs: K/ZDS/002839
Record Dates: First submitted 2016-05-16; First posted 2017-05-19 (Actual); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Surgical Complications From General Anesthesia; Cerebral Ischemia; Anesthesia; Reaction
Keywords: cerebral saturation; epidural anaesthesia; Near Infrared Spectroscopy (NIRS); Regional cerebral oxygen saturation
MeSH Terms: conditions — Brain Ischemia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- nirs: The cerebral oxymetry saturation was monitored continuously, using a non-invasive method. The cerebral saturation was monitored intraoperatively with near infrared spectroscopy (INVOS 4100; Somanetics Inc, Troy, MI). Data acquired from the device were automatically and continuously recorded in 10-second intervals throughout the anaesthesia. A lead for the cerebral saturation monitoring was placed on degreased skin on the patient's forehead, on the right side, some 1 cm over the eyebrow. The baseline value was determined before induction of anaesthesia. The following criteria were accepted as significant reduction of the cerebral oxygenation (saturation) value: reduction of the cerebral oxymetry by over 25% in relation to the baseline; the absolute value of cerebral oxymetry below 50%.
- cognitive function: Upon the day preceding the actual surgery, and again at 5 days after the surgery, the Mini Mental State Examination test was completed, with a view to assessing the chang-es in the patients' cognitive function. The difference between score in Mini Mental State Examination higher than 2 points defined a diagnosis of cognitive dysfunction.

SUMMARY:
Subsequent and non-randomised patients, adult patients qualified for major abdominal surgeries were enrolled

ELIGIBILITY:
Inclusion Criteria:

* scheduled for major abdominal surgery for at least 2 h
* under general anesthesia
* American Society of Anesthesiologists（ASA）physical status : II ~ III
* Age > 18

Exclusion Criteria:

* refuse of patients
* patient with results of test: "The Mini Mental State Examination"" less then 24 before operation
* neurosurgery history of patients

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: One hundred and one (101) subsequent and non-randomised patients, age between 35 and 84 years (mean 64±10) hospitalised at the 1st Department of General, Oncologic and Gastroenterologic Surgery of the UJ CM in Krakow, qualified for abdominal surgeries were enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2012-07; Primary Completion 2013-03 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
cerebral saturation | every 5 minutes throughout the surgery
  decreases in cerebral oxygen saturation (rSO2) during the surgery

SECONDARY OUTCOMES:
the Mini Mental State Examination test | Baseline, 4 day after surgery
  to assessing the changes in the patients' cognitive function

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Składzień, Ph.D, Study Chair — University Hospital in Cracow
Locations (1):
- University Hopital, Krakow, Małpololskie, Poland

IPD SHARING:
Plan to Share IPD: No
1. The day before the surgery will be performed basic blood tests (morphology, gas analysis) and test "Short Scale Mental State Examination."
  2. During the operation, in addition to standard monitoring the electrical activity of the heart, blood pressure and peripheral oxygen saturation levels, will be assessed non-invasively cerebral oximetry.
  3. When during general anesthesia bradycardia occurs, then half of the patients in this group will be set up into the esophagus electrode, which will provide the ability to route atrial pacing hemodynamically optimal heart rate (80 / min). However, in the second half of the patients at the time of the occurrence of bradycardia is given intravenously at a dose of atropine 0.5 mg.
  4. In about two hours after the surgery will be taken blood tests (morphology + gas analysis) to determine the potential impact of intraoperative bleeding changes oximetry.
  5. On postoperative day 5 will be repeated test "Short Scale Mental State Examination"